CLINICAL TRIAL: NCT04459585
Title: A Phase 1, Open-Label, Fixed Sequence Drug Interaction Study to Evaluate the Potential Intestinal Inhibitory Effect of Quizartinib on the Pharmacokinetics of a Pgp Substrate Dabigatran Etexilate in Healthy Subjects
Brief Title: A Study of the Effect of Quizartinib on the Pharmacokinetics of the P-gp Substrate Dabigatran Etexilate in Healthy Participants
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AC220-A-U104
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Healthy Subjects; Drug-drug Interaction; Pharmacokinetics; Quizartinib
Keywords: Healthy subjects; Drug-drug Interaction; Pharmacokinetics; Quizartinib; P-gp; Dabigatran Etexilate
MeSH Terms: interventions — Dabigatran; quizartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dabigatran + Quizartinib (Experimental): Participants who will receive a single oral dose of 150mg dabigatran etexilate on Day 1 of Period 1 and then will receive a single oral dose of 60mg quizartinib 2 hours prior to the administration of a single oral dose of 150mg dabigatran etexilate on the morning of Day 5 of Period 2.
  Interventions: Drug: Dabigatran Etexilate Mesylate; Drug: Quizartinib

INTERVENTIONS:
Drug: Dabigatran Etexilate Mesylate — Single oral 150 mg capsule dose
  Other Names: Pradaxa
Drug: Quizartinib — Single oral 60 mg dose of quizartinib administered as two 30 mg tablets (26.5 mg free base per tablet)

SUMMARY:
The purpose of this study is to investigate the one-way drug-drug interaction potential of quizartinib on dabigatran etexilate in healthy adult participants.

DETAILED DESCRIPTION:
This study will evaluate the potential intestinal inhibitory effect of quizartinib on the pharmacokinetics of a Pgp substrate dabigatran etexilate in healthy participants.

The hypothesis for this clinical study is that quizartinib, as a P-gp inhibitor, may increase the systemic exposure (measured by area under the concentration-time curve [AUC] and maximum concentration [Cmax]) of P-gp substrates that may be sensitive to intestinal P-gp inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 18 to 55 years of age (inclusive), with a body mass index (BMI) of 18 kg/m^2 to 32 kg/m^2 (inclusive) and with a minimum body weight of 45 kg at Screening.
* In females, documented surgical sterilization, postmenopausal status for at least 1 year (follicle stimulating hormone [FSH] > 40 million international (mIU)/mL serum at Screening), or agreement to use an approved form of contraception
* In males, agreement to avoid sperm donation for 6 months days after the dose of quizartinib
* Participants must agree to refrain from donation of blood from 56 days prior to Screening, plasma from 2 weeks prior to Screening, and platelets from 6 weeks prior to Screening.
* Liver function test results must be below the upper limit of normal. Hemoglobin levels must be ≥ 11.5 g/dL for female participants and ≥ 12.5 g/dL for male participants.
* All participants must be willing to refrain from consuming grapefruit/grapefruit juice, Seville oranges, and pomegranates/pomegranate juice 10 days before the dose of the study drug is given on Day 1 until end-of-study.

Exclusion Criteria:

* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including lab abnormality) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
* Laboratory results (serum chemistry, hematology, and urinalysis) outside the normal range, if considered clinically significant by the investigator. Estimated glomerular filtration rate (eGFR) < 90 mL/min at screening.
* Women who are pregnant or breastfeeding
* Use of any drugs or substances known to be inhibitors or inducers of CYP3A4/5 within 28 days from the first dose or 5 half-lives, if known, of the drugs or substances, whichever is greater, prior to quizartinib administration and during the study.
* Receipt of any prescribed or over-the-counter (OTC) systemic, herbal (including St John's wort), or topical medication within 14 days of quizartinib administration, or any expectation of requiring use of such medication while participating in the study is prohibited.
* Presence or history of clinically severe adverse reaction to any drug
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (with the exception of appendectomy, hernia repair, and/or cholecystectomy)
* A positive drugs of abuse screen from a urine ethanol test (unless the drug is medically prescribed by a licensed health care provider) or alcohol breath test at Screening or at Check-in on Day -1 or a participant who will not agree to smoke ≤10 cigarettes or equivalent per day from Screening up to Enrollment, and is unable to be restricted to ≤5 cigarettes per day and for 6 hours post dose during their period of residence in the clinical unit
* Concomitant use of medications known to affect the elimination of serum creatinine (e.g., trimethoprim or cimetidine) and inhibitors of renal tubular secretion (eg, probenecid) within 14 days or 5 half-lives, if known, of the drugs, whichever is greater, prior to quizartinib administration
* History or presence of an abnormal electrocardiogram (ECG), which, in the investigator's opinion, is clinically significant and/or a QT interval corrected for heart rate using Fridericia's formula >450 milliseconds (ms) at Screening.
* Use of drugs with a risk of QT interval prolongation or torsade de pointes within 14 days of Day -1 (or 5 drug half-lives, if 5 drug half-lives are expected to exceed 14 days)
* Consumption of alcohol- and caffeine-containing beverages within 72 hours prior to check-in and during confinement
* Positive serology for hepatitis B surface antigen (HBsAg) and hepatitis C virus [HCV] (healthy participants), hepatitis A virus (HAV) immunoglobulin M, or anti-human immunodeficiency virus (HIV) Type 1 and Type 2 (all subjects)
* Current enrollment in or have not yet completed at least 30 days or 5 elimination half-lives, whichever is longer, since receiving an investigational device or product, or receipt of other investigational agents within 30 days of quizartinib

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 20 participants who met all inclusion criteria and no exclusion criteria were enrolled from 28 Aug 2020 to 20 Oct 2020 at 1 clinic in the United States.
Pre-assignment Details: This study consisted of two treatment periods. Following a Screening Period of 21 days, eligible participants received only dabigatran etexilate (Reference Treatment) on Day 1 of Period 1 followed by quizartinib and dabigatran etexilate administration (Test Treatment) on Day 5 of Period 2.
Groups:
- Dabigatran Etexilate/Dabigatran Etexilate + Quizartinib: Participants who received a single oral dose of 150mg dabigatran etexilate on Day 1 of Period 1 and then received a single oral dose of 60mg quizartinib 2 hours prior to the administration of a single oral dose of 150mg dabigatran etexilate on the morning of Day 5 of Period 2.
Period: Period 1 (Day 1 to Day 5)
Arm/Group | Dabigatran Etexilate/Dabigatran Etexilate + Quizartinib
Started | 20
Completed | 20
Not Completed | 0
Period: Period 2 (Day 5 to Day 12)
Arm/Group | Dabigatran Etexilate/Dabigatran Etexilate + Quizartinib
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed using the Safety Analysis Set.
Arm/Group | Dabigatran Etexilate/Dabigatran Etexilate + Quizartinib
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Total Dabigatran and of Free Dabigatran Following a Single Dose in Participants Without and With Concomitant Quizartinib
Description: Maximum Plasma Concentration (Cmax) is defined as the maximum observed plasma concentration and was calculated using non-compartmental analysis.
Time Frame: Period 1 Day 1 (Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60 and 72 hours post-dose) and Period 2 Day 5 (pre-dose and 1, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 14, 26, 38, 50, 62, and 74 hours post-dose)
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Period 1: Dabigatran Etexilate: Participants who received a single oral dose of 150mg dabigatran etexilate on Day 1 of Period 1.
- Period 2: Dabigatran Etexilate + Quizartinib: Participants who received a single oral dose of 60mg quizartinib 2 hours prior to the administration of a single oral dose of 150mg dabigatran etexilate on Day 5 of Period 2.
Arm/Group | Period 1: Dabigatran Etexilate | Period 2: Dabigatran Etexilate + Quizartinib
Number analyzed (Participants) | 20 | 20
ng/mL
  Total Dabigatran | 192 (94.5) | 239 (141)
  Free Dabigatran | 159 (82.2) | 201 (127)
Statistical Analysis 1: Comparison: Period 1: Dabigatran Etexilate vs Period 2: Dabigatran Etexilate + Quizartinib; Statistical comparison was analyzed for Total Dabigatran; Test type: Other — Least squares (LS) means were calculated from an analysis of variance (ANOVA) model on log-transformed scale. The LS means for each treatment were back transformed from the log scale to provide estimates of the geometric means (GMS). The ratio (%) of GMS was calculated and 90% Confidence Intervals (CIs) for the ratio (%) of GMS were presented; Ratio (%) of Geometric LS Mean = 111.88, 90% CI 2-sided [77.57 to 161.35] — For the comparison, the Dabigatran Etexilate + Quizartinib (Period 2) represents the numerator and Dabigatran Etexilate (Period 1) represents the denominator
Statistical Analysis 2: Comparison: Period 1: Dabigatran Etexilate vs Period 2: Dabigatran Etexilate + Quizartinib; Statistical comparison was analyzed for Free Dabigatran; Test type: Other — Least squares (LS) means were calculated from an analysis of variance (ANOVA) model on log-transformed scale. The LS means for each treatment were back transformed from the log scale to provide estimates of the geometric means (GMS). The ratio (%) of GMS was calculated and 90% CIs for the ratio (%) of GMS were presented; Ratio (%) of Geometric LS Mean = 112.98, 90% CI 2-sided [77.20 to 165.34] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve up to the Last Quantifiable Concentration Post-Dose (AUClast) of Total Dabigatran and of Free Dabigatran Following a Single Dose in Participants Without and With Concomitant Quizartinib
Description: Area Under the Plasma Concentration-Time Curve up to the Last Quantifiable Concentration Post-Dose (AUClast) is defined as AUC from time 0 to the last measurable concentration, as calculated by the linear up-log down trapezoidal method and was calculated using non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Period 1: Dabigatran Etexilate | Period 2: Dabigatran Etexilate + Quizartinib
Number analyzed (Participants) | 20 | 20
ng*h/mL
  Total Dabigatran | 1720 (870) | 2100 (1280)
  Free Dabigatran | 1390 (736) | 1710 (1100)
Statistical Analysis 1: Comparison: Period 1: Dabigatran Etexilate vs Period 2: Dabigatran Etexilate + Quizartinib; Statistical comparison was analyzed for Total Dabigatran; Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (%) of Geometric LS Mean = 111.37, 90% CI 2-sided [78.51 to 157.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Period 1: Dabigatran Etexilate vs Period 2: Dabigatran Etexilate + Quizartinib; Statistical comparison was analyzed for Free Dabigatran; Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (%) of Geometric LS Mean = 111.08, 90% CI 2-sided [77.35 to 159.51] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Area Under the Plasma Concentration-Time Curve up to Infinity (AUCinf) of Total Dabigatran and of Free Dabigatran Following a Single Dose in Participants Without and With Concomitant Quizartinib
Description: Area Under the Plasma Concentration-Time Curve up to Infinity (AUCinf) is defined as area under the plasma concentration-time curve from the time of dosing extrapolated to infinity and was calculated using non-compartmental analysis.
Time Frame: as for outcome 1
Population: The pharmacokinetic parameter of Area Under the Plasma Concentration-Time Curve up to Infinity was assessed using the Pharmacokinetic Analysis Set except for 1 participant that did not meet the protocol inclusion criteria for this analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Period 1: Dabigatran Etexilate | Period 2: Dabigatran Etexilate + Quizartinib
Number analyzed (Participants) | 20 | 20
ng*h/mL
  Total Dabigatran: number analyzed (Participants) | 19 | 20
  Total Dabigatran | 1740 (902) | 2140 (1280)
  Free Dabigatran: number analyzed (Participants) | 19 | 20
  Free Dabigatran | 1420 (760) | 1730 (1100)
Statistical Analysis 1: Comparison: Period 1: Dabigatran Etexilate vs Period 2: Dabigatran Etexilate + Quizartinib; Statistical comparison was analyzed for Total Dabigatran; Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (%) of Geometric LS Mean = 112.97, 90% CI 2-sided [79.38 to 160.79] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Period 1: Dabigatran Etexilate vs Period 2: Dabigatran Etexilate + Quizartinib; Statistical comparison was analyzed for Free Dabigatran; Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (%) of Geometric LS Mean = 110.72, 90% CI 2-sided [76.77 to 159.68] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of Total Dabigatran and of Free Dabigatran Following a Single Dose in Participants Without and With Concomitant Quizartinib
Description: Time of Maximum Plasma Concentration (Tmax) is defined as time of maximum observed plasma concentration and was calculated using non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Period 1: Dabigatran Etexilate | Period 2: Dabigatran Etexilate + Quizartinib
Number analyzed (Participants) | 20 | 20
hours
  Total Dabigatran | 2.0 [1.5 to 3.1] | 2.0 [1.5 to 4.0]
  Free Dabigatran | 2.0 [1.5 to 4.0] | 2.0 [1.5 to 4.0]

5. Secondary Outcome: Terminal Elimination Half-Life (T1/2) of Total Dabigatran and of Free Dabigatran Following a Single Dose in Participants Without and With Concomitant Quizartinib
Description: Terminal Elimination Half-Life (T1/2) is defined as terminal elimination half-life and was calculated using non-compartmental analysis.
Time Frame: as for outcome 1
Population: The pharmacokinetic parameter of Terminal Elimination Half-Life was assessed using the Pharmacokinetic Analysis Set except for 1 participant that did not meet the protocol inclusion criteria for this analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Period 1: Dabigatran Etexilate | Period 2: Dabigatran Etexilate + Quizartinib
Number analyzed (Participants) | 20 | 20
hours
  Total Dabigatran: number analyzed (Participants) | 19 | 20
  Total Dabigatran | 15.4 (4.4) | 18.1 (17.0)
  Free Dabigatran: number analyzed (Participants) | 19 | 20
  Free Dabigatran | 14.2 (4.2) | 14.1 (6.6)

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Quizartinib and the Metabolite ACC886 Following Single Dose of Dabigatran With Quizartinib in Participants
Description: Maximum Plasma Concentration (Cmax) is defined as the maximum observed plasma concentration and was calculated using non-compartmental analysis. Cmax was assessed for Quizartinib and Metabolite AC886.
Time Frame: Period 2 Day 5 (Pre-dose and 1, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 14, 26, 38, 50, 62, and 74 hours post-dose)
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Median (Standard Deviation); unit: ng/mL
Arm/Group | Period 2: Dabigatran Etexilate + Quizartinib
Number analyzed (Participants) | 20
ng/mL
  Quizartinib | 250 (50.8)
  AC886 | 25.7 (8.71)

7. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of Quizartinib and the Metabolite ACC886 Following Single Dose of Dabigatran With Quizartinib in Participants
Description: Time of Maximum Plasma Concentration (Tmax) is defined as time of maximum observed plasma concentration and was calculated using non-compartmental analysis. Tmax was assessed for Quizartinib and Metabolite AC886.
Time Frame: Period 2 Day 5 (Pre-dose and 1, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 14, 26, 38, 50, 62, and 74 hours post-dose)
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Period 2: Dabigatran Etexilate + Quizartinib
Number analyzed (Participants) | 20
hours
  Quizartinib | 3.0 [2.5 to 6.0]
  AC886 | 8.0 [3.5 to 26.1]

8. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to 74 Hours (AUClast,74) of Quizartinib and the Metabolite ACC886 Following Single Dose of Dabigatran With Quizartinib in Participants
Description: Area Under the Plasma Concentration-Time Curve From Time 0 to 74 Hours (AUClast,74) is defined as area under the plasma concentration-time curve to the last quantifiable concentration post dose at 74 hours and was calculated using non-compartmental analysis. AUClast,74 was assessed for Quizartinib and Metabolite AC886.
Time Frame: Period 2 Day 5 (Pre-dose and 1, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 14, 26, 38, 50, 62, and 74 hours post-dose)
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Period 2: Dabigatran Etexilate + Quizartinib
Number analyzed (Participants) | 20
ng*h/mL
  Quizartinib | 9390 (1660)
  AC886 | 1350 (495)

9. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAE) Relatedness to Study Medication Following Single Dose of Dabigatran Without and With Quizartinib in Participants
Description: A Treatment-Emergent Adverse Events (TEAE) is defined as any event not present prior to the initiation of the drug treatment of the drug treatment or any event already present that worsens in either intensity or frequency following exposure to the drug treatment. Number of any TEAE that is related and unrelated to study medication is presented.
Time Frame: Up to 2 months
Population: TEAEs were assessed using the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Dabigatran Etexilate | Period 2: Dabigatran Etexilate + Quizartinib
Number analyzed (Participants) | 20 | 20
Participants
  Related | 0 | 2
  Unrelated | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of signing the informed consent form up to 30 days after last dose, up to 2 months.
Description: Adverse events were defined as any untoward, unfavorable, unintended medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. All-cause mortality includes all deaths that occurred during the study and within the 30 days after the last dose of the study drug.
Arm/Group | Period 1: Dabigatran Etexilate | Period 2: Dabigatran Etexilate + Quizartinib
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 3/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: Dabigatran Etexilate (N=20) | Period 2: Dabigatran Etexilate + Quizartinib (N=20)
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT04459585/Prot_SAP_000.pdf